CLINICAL TRIAL: NCT02987699
Title: Phase II Study of Hepatic Arterial Infusion Chemotherapy Using Oxaliplatin,Leucovorin and 5-Fluorouracil
Brief Title: Phase II Study of HAIC Using Cisplatin,Leucovorin and 5-Fluorouracil
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unique Protocol ID: HCC-S026
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: HepatoCellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy; optimal dose
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full Dosage (Experimental): Full Dosage Chemotherapy regimen administered by HAI
  Interventions: Drug: 5-Fu, oxaliplatin , leucovorin
- Low Dosage of 5-Fu (Experimental): Low Dose of 5-Fu Chemotherapy regimen administered by HAI
  Interventions: Drug: 5-Fu, oxaliplatin , leucovorin
- Low Dosage of oxaliplatin (Experimental): Low Dose of oxaliplatin Chemotherapy regimen administered by HAI
  Interventions: Drug: 5-Fu, oxaliplatin , leucovorin

INTERVENTIONS:
Drug: 5-Fu, oxaliplatin , leucovorin — Drug: 5-Fu, oxaliplatin and regular dose of leucovorin Regimen: (1) 5-Fu: 2800 mg/m2 (2) oxaliplatin: 135 mg/m2 (3) leucovorin: 400mg/m2
  Other Names: Full dose Folfox
  Arms: Full Dosage
Drug: 5-Fu, oxaliplatin , leucovorin — Drug: 5-Fu, oxaliplatin and regular dosage of leucovorin Regimen: (1) 5-Fu: 1400 mg/m2 (2) oxaliplatin: 135 mg/m2 (3) leucovorin: 400mg/m2
  Other Names: Low dose 5-Fu Folfox
  Arms: Low Dosage of 5-Fu
Drug: 5-Fu, oxaliplatin , leucovorin — Drug: 5-Fu, oxaliplatin and regular dosage of leucovorin Regimen: (1) 5-Fu: 2800 mg/m2 (2) oxaliplatin: 85 mg/m2 (3) leucovorin: 400mg/m2
  Other Names: Low dose oxaliplatin Folfox
  Arms: Low Dosage of oxaliplatin

SUMMARY:
The purpose of this phase II study is to determine the recommended dose, as well as the safety and efficacy of the combination of oxaliplatin, leucovorin and 5-Fu introduced by hepatic arterial infusion chemotherapy (HAIC) in patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The results of our preliminary pilot study suggested that the combination of oxaliplatin, leucovorin and 5-Fu introduced by hepatic arterial infusion chemotherapy (HAIC) may improve the survivals for advanced stage HCC. Thus, the investigators carried out this prospective randomized control study to determine the recommended dose as well as the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL) Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.

diagnosed with major or main portal vein invasion (Vp3 or Vp4) KPS≥70； with no previous treatment No Cirrhosis or cirrhotic status of Child-Pugh class A only Not amendable to surgical resection ,local ablative therapy and any other cured treatment.

The following laboratory parameters:

Platelet count ≥ 75,000/µL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3 Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy Known history of HIV History of organ allograft Known or suspected allergy to the investigational agents or any agent given in association with this trial.

Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy Evidence of bleeding diathesis. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug Serious non-healing wound, ulcer, or bone fracture Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 3 Months
  Tumor response evaluated by postoperative CT/MRI scan according to RECIST criteria.

SECONDARY OUTCOMES:
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03
Number of of Patients developed Adverse Events | 30 days
  Number of of patients who developed adverse event. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, Doctor, Principal Investigator — The Department of Hepatobiliary Pancreatic Oncology of Sun Yat-sen University Cancer Center
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794